CLINICAL TRIAL: NCT01649401
Title: Efficacy of the PARI LC Sprint Sp Nebulizer for Acute Asthma Attack in Hospitalized Children Less Than 36 Months of Age
Acronym: LC SPRINT Sp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2012/LG-02; 2012-A00629-34 (Other: RCB)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
Keywords: nebulizer; PARI LC Spring SP
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard nubulizer (Active Comparator): Nebulizer sessions for the patients in this arm will be administerd using our "standard" nebulizer: Micro Mist, ref 41894, Hudson RCI, distributed by Téléflex Médical.
  Interventions: Device: Standard nebulizer
- Experimental nebulizer (Experimental): Nebulizer sessions for the patients in this arm will be administerd using the PARI LC Sprint Sp nebulizer.
  Manufacturer: PARI GmbH Germany
  Interventions: Device: PARI LC Sprint Sp nebulizer

INTERVENTIONS:
Device: Standard nebulizer — Nebulizer sessions for the patients will be administerd using our "standard" nebulizer: Micro Mist, ref 41894, Hudson RCI, distributed by Téléflex Médical.
  Other Names: Micro Mist Nebulizer
  Arms: Standard nubulizer
Device: PARI LC Sprint Sp nebulizer — Nebulizer sessions for the patients will be administerd using the PARI LC Sprint Sp nebulizer.
  Manufacturer: PARI GmbH Germany
  Arms: Experimental nebulizer

SUMMARY:
The main objective of this study is to determine whether the use of the PARI LC Sprint Sp nebulizer in the treatment of asthma in children under 36 months reduces the duration of hospitalization.

DETAILED DESCRIPTION:
The secondary objectives of this study are to evaluate whether the use of the LC Sprint Sp Nebulizer results in:

A-shortened duration of oxygen-dependence.

B-reduced side effects by assessing the patient's heart rate before and 30 minutes after the first aerosol and noting the occurrence of desaturation <90% during the nebulisation sessions.

C-increased acceptance of the aerosol, measured via a questionnaire given to the patient's parents at the end of hospitalization (a single questionnaire will be completed by either parent or both parents).

D-shortened length of stay based on the following discharge criteria: observation of a respiratory severity score ≤ 2 (Clinical Asthma Score (CAS)) for at least 12 consecutive hours and a transcutaneous oxygen saturation (SpO2)> 94% when awake or > 91% during sleep.

ELIGIBILITY:
Inclusion Criteria:

* The parent or legal representative must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has an attack of moderate to severe asthma (at least the third episode of wheezing dyspnea since birth) requiring hospitalization defined by the following criteria:
* requires oxygen: SpO2 <92% on room air (if CAS ≤ 4/10)

  * And / or CAS> 4/10 (after 3 attempted nebulized salbutamol sessions over 1 hour of emergency care).

Exclusion Criteria:

* The patient is participating in another study
* The patients has already been included in this study a previous time
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The parent or legal representative refuses to sign the consent
* It is impossible to correctly inform the parent or legal representative
* The patient has a contra indication for a treatement used in this study
* Patient was born at < 34 weeks of pregnancy or bronchdysplasic
* First or second episode of bronchiolitis
* Asthma attack with CAS score ≤ 4/10 or inpatient basis for a non-breathing related motive.
* Acute severe Asthma attack: hypercapnia, impaired consciousness, need for hospitalization in intensive care, need for mechanical ventilation, need for salbutamol IV
* Patient with known congenital heart disease
* Patient with chronic respiratory disease other than asthma
* Patient with encephalopathy
* Patient with known immune deficiency
* CAS ≤ 2 and transcutaneous oxygen saturation (SpO2)> 94% when awake or > 91% when asleep for at least 12h

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2012-12; Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | hospital discharge (maximum of 10 days)
  The length of hospitalization in days

SECONDARY OUTCOMES:
Duration of oxygen therapy | Day 0
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Heart rate before the first nebulisation session | Day 0
  Heart rate before the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 0
  Heart rate 30 minutes after the first nebulisation session (bpm)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 0
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
Duration of oxygen therapy | Day 1
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 2
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 3
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 4
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 5
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 6
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 7
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 8
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 9
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Duration of oxygen therapy | Day 10
  Duration of oxygen therapy (necessary to return to a saturation of > 91% when sleep, or > 94% when awake); measured in hours
Heart rate before the first nebulisation session | Day 1
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 2
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 3
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 4
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 5
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 6
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 7
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 8
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 9
  Heart rate before the first nebulisation session (bpm)
Heart rate before the first nebulisation session | Day 10
  Heart rate before the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 1
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 2
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 3
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 4
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 5
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 6
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 7
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 8
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 9
  Heart rate 30 minutes after the first nebulisation session (bpm)
Heart rate 30 minutes after the first nebulisation session | Day 10
  Heart rate 30 minutes after the first nebulisation session (bpm)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 1
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 2
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 3
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 4
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 5
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 6
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 7
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 8
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 9
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
SpO2 saturation less thant 90% during or after nebulisation session? | Day 10
  Does the SpO2 saturation drop to less thant 90% during or after nebulisation session? (up to 30 minutes after the session; yes/no)
Parent estimated tolerance | Hospital discharge (maximum 10 days)
  A visual analog scale is used to evaluate how parents estimate aerosol tolerance.
Length of hospitalization according to discharge criteria | Hospital discharge (maximum 10 days)
  length of stay based on the following discharge criteria: observation of a respiratory severity score ≤ 2 (Clinical Asthma Score CAS) for at least 12 consecutive hours and a transcutaneous oxygen saturation (SpO2)> 94% when awake or > 91% during sleep

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Gilton-Bott, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France